CLINICAL TRIAL: NCT06052137
Title: Open Label - Personalized Therapeutic Neuromodulation for Anhedonic Depression
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, David Spiegel, Professor, Psychiatry and Behavioral Sciences, Stanford School of Medicine, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 71771
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Treatment Resistant Depression
Keywords: transcranial magnetic stimulation; theta burst
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active TBS-DLPFC (Active Comparator): The active group will receive theta-burst TMS DLPFC stimulation.
  Interventions: Device: Active TBS-DLPFC
- Active TBS-DMPFC (Active Comparator): The active group will receive theta-burst TMS DMPFC stimulation.
  Interventions: Device: TBS-DMPFC

INTERVENTIONS:
Device: Active TBS-DLPFC — Participants will receive intermittent TBS to left DLPFC. The L-DLPFC will be targeted utilizing the Localite neuronavigation system. Stimulation intensity will be standardized at 90% of RMT and adjusted to the skull to cortical surface distance (see Nahas 2004).
  Stimulation will be delivered to the L-DLPFC using a MagPro TMS system (MagVenture, Denmark).
  Arms: Active TBS-DLPFC
Device: TBS-DMPFC — Participants will receive intermittent TBS to DMPFC. The DMPFC will be targeted utilizing the Localite neuronavigation system. Stimulation intensity will be standardized at 90% of RMT and adjusted to the skull to cortical surface distance (see Nahas 2004).
  Stimulation will be delivered to the DMPFC using a MagPro TMS system (MagVenture, Denmark).
  Arms: Active TBS-DMPFC

SUMMARY:
This study will investigate the anti-anhedonic efficacy of a novel neurostimulation strategy termed accelerated intermittent theta burst stimulation (aiTBS) in participants with treatment resistant depression (TRD).

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) is an established therapy for treatment-resistant depression. The approved method for treatment is 10Hz stimulation for 40 min over the left dorsolateral prefrontal cortex (L-DLPFC). This methodology has been effective in real world situations. The limitations of this approach include the duration of the treatment (approximately 40 minutes per treatment session, 5 days per week, for 4-8 weeks). Recently, the investigators have pursued modifying the treatment parameters to reduce treatment times with an accelerated treatment paradigm. This study aims to further study the accelerated protocol and examine changes in neuroimaging biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, between the ages of 18 and 80 at the time of screening.
2. Able to read, understand, and provide written, dated informed consent prior to screening. Proficiency in English sufficient to complete questionnaires / follow instructions during fMRI assessments and aiTBS interventions. Stated willingness to comply with all study procedures, including availability for the duration of the study, and to communicate with study personnel about adverse events and other clinically important information.
3. Currently diagnosed with Major Depressive Disorder (MDD) and meets criteria for a Major Depressive Episode, according to the criteria defined in the Diagnosis and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision (DSM-5).
4. MADRS score of ≥20 at screening (Visit 1).
5. TMS naive for one of the following areas: DLPCF or DMPFC
6. The dose of the primary antidepressant medication (if applicable) must be stable for 6 weeks prior to baseline, and participant must agree to continue at this dose throughout the study period.
7. In good general health, as evidenced by medical history.
8. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation.
9. Agreement to adhere to Lifestyle Considerations throughout study duration.

Lifestyle Considerations:

* Abstain from becoming pregnant from the screening visit (Visit 1) until after the final study visit (Visit 10).
* Abstain from caffeine- or xanthine-containing products (e.g., coffee, tea, cola drinks, and chocolate) for 3 hours before the start of each dosing session until after the final TMS session.
* Abstain from alcohol for 24 hours before the start of each dosing session until after collection of the final MRI.
* Participants who use tobacco products will be instructed that use of cigarettes will not be allowed during the study.

Exclusion Criteria:

1. Pregnancy
2. History of or current psychotic disorder or bipolar disorder
3. Severe borderline personality disorder.
4. Diagnosis of Intellectual Disability or Autism Spectrum Disorder
5. Primary psychiatric condition other than MDD requiring treatment except stable comorbid anxiety disorder
6. Current moderate or severe substance use disorder or demonstrating signs of acute substance withdrawal
7. Urine screening test positive for illicit substances
8. Acute suicide risk based on clinical judgement or a suicide attempt (as defined by the C-SSRS) within the past one year
9. Any history of ECT (greater than 8 sessions) without meeting responder criteria
10. Recent (within 4 weeks of any clinical effect) or concurrent use of rapid acting antidepressant agent (i.e., ketamine or a course of ECT)
11. History of significant neurologic disease, including dementia, Parkinson's or Huntington's disease, brain tumor, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma
12. Untreated or insufficiently treated endocrine disorder.
13. Contraindication to receiving rTMS (e.g., metal in head, history of seizure, known brain lesion)
14. Contraindication to MRI (ferromagnetic metal in their body)
15. Treatment with an investigational drug or other intervention within the study period
16. Depth-adjusted aiTBS treatment dose > 65% maximum stimulator output (MSO)
17. Unstable symptoms between screening and baseline as defined by a ≥ 30% change in MADRS score.
18. Any other condition deemed by the PD to interfere with the study or increase risk to the participant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-12-19 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Change in clinician-administered MADRS from Baseline to Week 1 post-treatment-initiation | Baseline, 1-week post-treatment-initiation
  The Montgomery-Asberg Depression Rating Scale (MADRS) is a 10-item clinician-administered scale, designed to be particularly sensitive to antidepressant treatment effects in patients with major depression. Score range of 0-60. A higher score is indicative of more depression.

CONTACTS AND LOCATIONS:
Overall Officials: David Spiegel, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No